CLINICAL TRIAL: NCT05373095
Title: Strengthening the Continuity of HIV Care in Tanzania With Economic Support: Phase II
Brief Title: Rudi Kundini, Pamoja Kundini
Acronym: RKPK: Phase II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Health for a Prosperous Nation (Other); Rasello (Industry); Management and Development for Health (Unknown); Ministry of Health, Tanzania (Other Government); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R01MH125746 - Phase II; R01MH125746 (NIH)
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: Tanzania; Conditional Cash Transfers; People Living With HIV; Machine Learning
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Laboratory staff analyzing viral load samples will be blind to intervention/control attribution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Adherence Counseling (PKC) and Conditional Cash Transfers (Experimental): Eligible and consenting participants randomized to the intervention arm will receive the same standard HIV clinical services according Tanzania's National Guidelines for the Management of HIV as the comparison arm, which includes provision of three, once-monthly, 60-minute nurse-led individual, enhanced adherence counseling sessions adapted for study purposes (PKC sessions). Counseling focuses on the meaning of viral loads and supportive, non-judgmental strategies for adherence and visit attendance. A minimum of three sessions are required. In addition to enhanced adherence counseling, intervention participants will receive the offer of a cash transfer paired with attendance at each of the three enhanced adherence counseling sessions. The first payment will occur at enrollment; the next two cash transfers are payable upon visit attendance and attendance of the two remaining enhanced adherence counseling sessions.
  Interventions: Behavioral: PKC (adapted adherence counseling) and Conditional Cash Transfers
- Enhanced Adherence Counseling only for those who qualify (No Intervention): Eligible and consenting participants randomized to the control arm will receive standard of care HIV clinical services according to Tanzania's National Guidelines for the Management of HIV. For those who meet clinic eligibility criteria for enhanced adherence counseling, this includes the standard provision of three, once-monthly, 60-minute nurse-led individual, enhanced adherence counseling sessions, starting on the day of a detectable viral load result and for two months after. Counseling focuses on the meaning of viral loads and supportive, non-judgmental strategies for adherence and visit attendance. A minimum of three sessions are required.

INTERVENTIONS:
Behavioral: PKC (adapted adherence counseling) and Conditional Cash Transfers — The intervention includes up to 3 cash transfers of 22,500 Tanzanian Shillings (~$10) paired with attendance at each of the three adapted enhanced adherence counseling sessions (PKC sessions). The first cash transfer will occur at enrollment; the next two cash transfers are payable upon visit attendance and attendance of the two remaining PKC sessions. The cash transfers will include extra funds for transaction fees, typically <$1.
  Arms: Adapted Adherence Counseling (PKC) and Conditional Cash Transfers

SUMMARY:
This protocol describes an individually randomized trial that will include adult people living with HIV (PLHIV) currently receiving HIV care at one of two participating health facilities and identified as high risk for disengagement from care by a machine learning algorithm. Participants randomized to the control arm will receive standard of care HIV clinical services according to Tanzania's National Guidelines for the management of HIV. For those who meet clinic eligibility criteria for enhanced adherence counseling, which at the included study sites is when client's viral load reaches a detectable level (>1000 copies/ml), this includes the standard provision of three, once-monthly, 60-minute nurse-led individual, enhanced adherence counseling sessions, starting on the day of the result and for two months after. Intervention arm participants will receive the same standard HIV care services plus the offer of a cash transfer paired with visit attendance and attendance at each of the three adapted enhanced adherence counseling sessions (referred to as PKC sessions).

DETAILED DESCRIPTION:
This protocol describes a 2-armed parallel individually randomized controlled trial for which 692 PLHIV who meet eligibility criteria, are currently accessing care at a participating health facility (Katoro Health Center, Geita Town Council Hospital, Geita Regional Referral Hospital, or Nyankumbu Health Center), and have provided informed consent to be part of the study will be randomized in a 1:1 ratio (n=346 PLHIV in each arm), stratified by site, to the control or intervention group. The investigators will use machine learning to finalize a predictive model based on routinely collected medical and pharmacy record data to identify and recruit PLHIV for participation at participating facilities who are at high-risk for disengaging from HIV care.

Eligible and consenting participants randomized to the control arm will receive standard of care HIV clinical services according to Tanzania's National Guidelines for the Management of HIV. Criteria for enrollment into enhanced adherence counseling sessions includes when client's viral load reaches a detectable level (>1000 copies/ml). Enhanced adherence counseling includes the standard provision of three, once-monthly, 60-minute nurse-led individual, enhanced adherence counseling sessions, starting on the day of the result and for two months after. Counseling focuses on the meaning of viral loads and supportive, non-judgmental strategies for adherence and visit attendance. Sessions are conducted in an individual, 1:1 setting with a trained counselor who is on the clinical staff, or in a group setting with a trained counselor who is on the clinical staff. A minimum of three sessions are required. Eligible and consenting participants randomized to the intervention arm will receive the same standard HIV care services plus the offer of a cash transfer paired with visit attendance and attendance at each of the three adapted enhanced adherence counseling sessions (PKC sessions). The first payment will occur at enrollment; the next two cash transfers are payable upon visit attendance and attendance of the two remaining enhanced adherence counseling sessions. Due to the nature of the intervention, participants will not be blinded to intervention assignment. The primary endpoint is viral load suppression (<1000 copies/ml) at 12 months following study enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. PLHIV on ART;
2. Age 18 years or older;
3. Phone ownership OR consistent phone access;
4. Not already enrolled in/currently attending enhanced adherence counseling sessions at the facility
5. Living in Geita Region and intends to receive care at a study facility for the next 12 months;
6. Classified as "high-risk" for loss to follow-up (LTFU) from HIV care, and
7. Provides written informed consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
12-Month Viral Suppression | 12 months
  The proportion of people living with HIV (PLHIV) and on ART with suppressed HIV viral load ( <1000 copies/ml) at 12 months after study enrollment.

SECONDARY OUTCOMES:
6-month retention in care | 6 months
  The proportion of people living with HIV (PLHIV) on ART at 6 months after study enrollment (PEPFAR considers those not retained on ART to include those who died, disengaged from care, stopped ART, or had no evidence of care for ≥28 days after a missed visit. Participants not found after exhaustive tracing efforts to rule out silent transfers will be classified as not retained on ART)
12-month retention in care | 12 months
  The proportion of people living with HIV (PLHIV) on ART at 12 months after study enrollment (PEPFAR considers those not retained on ART to include those who died, disengaged from care, stopped ART, or had no evidence of care for ≥28 days after a missed visit. Participants not found after exhaustive tracing efforts to rule out silent transfers will be classified as not retained on ART)
12-month durable viral load | 12 months
  Proportion with durable HIV viral suppression 12 months after enrollment: at least 2 viral load measurements taken from up to 6 months prior to study enrollment and up to and including 12 months following study enrollment and all are undetectable (<1000 copies/ml) will have met criteria for durable viral suppression at 12 months.
12-month Appointment Attendance | 12 months
  The proportion of scheduled visits that were completed during the 0-12 month period
6-month Appointment Attendance | 6 months
  The proportion of scheduled visits that were completed during the 0-6 month period
12-month Mortality | 12 months
  The cumulative incidence of mortality at 12 months after study enrollment
6-month Predictive value positive (PVP) of machine learning algorithm | 6 months
  Predictive value positive (PVP) of the machine learning algorithm in identifying PLHIV at-risk of disengagement from HIV care within 6 months
12-month Predictive value positive (PVP) of machine learning algorithm | 12 months
  Predictive value positive (PVP) of the machine learning algorithm in identifying PLHIV at-risk of disengagement from HIV care within 12 months
6-month PVP of routine clinical criteria | 6 months
  PVP of the routine clinical criteria (i.e. recent missed visit or detectable viral load, >1000 copies/ml) for identifying PLHIV at-risk of disengagement from HIV care within 6 months
12-month PVP of routine clinical criteria | 12 months
  PVP of the routine clinical criteria (i.e. recent missed visit or detectable viral load, >1000 copies/ml) for identifying PLHIV at-risk of disengagement from HIV care within 12 months
6-month Predictive value negative (PVN) of the machine learning algorithm | 6 months
  Predictive value negative (PVN) of the machine learning algorithm in identifying PLHIV not at-risk of disengagement from HIV care within 6 months
12-month PVN of the machine learning algorithm | 12 months
  PVN of the machine learning algorithm in identifying PLHIV not at-risk of disengagement from HIV care within 12 months
6-month PVN of routine clinical criteria | 6 months
  PVN of the routine clinical criteria for identifying PLHIV not at-risk of disengagement from HIV care within 6 months
12-month PVN of routine clinical criteria | 12 months
  PVN of the routine clinical criteria for identifying PLHIV not at-risk of disengagement from HIV care within 12 months
Enhanced Adherence Counseling Session Attendance | 6 months
  Proportion of enhanced adherence counseling sessions completed among sessions scheduled
Viral Suppression with enhanced adherence counseling completion | 6 months
  Proportion with HIV viral suppression after completion of enhanced adherence counseling sessions
6-Month Viral Suppression (<1000 copies/ml) | 6 months
  The proportion of people living with HIV (PLHIV) and on ART with suppressed HIV viral load ( <1000 copies/ml) at 6 months after study enrollment.
6-Month Viral Suppression (<50 copies/ml) | 6 months
  The proportion of people living with HIV (PLHIV) and on ART with suppressed HIV viral load ( <50 copies/ml) at 6 months after study enrollment.
12-Month Viral Suppression (<50 copies/ml) | 12 months
  The proportion of people living with HIV (PLHIV) and on ART with suppressed HIV viral load ( <50 copies/ml) at 12 months after study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Jingshen Wang, PhD, Principal Investigator — University of California, Berkeley
Locations (4):
- Tanzania (4):
  - Geita Regional Referral Hospital, Geita
  - Geita Town Council Hospital, Geita
  - Nyankumbu Health Center, Geita
  - Katoro Health Center, Katoro

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Provided upon request

REFERENCES:
- [Derived] Kadota JL, Packel LJ, Mlowe M, Ulenga N, Mwenda N, Njau PF, Dow WH, Wang J, Sabasaba A, McCoy SI. Rudi Kundini, Pamoja Kundini (RKPK): study protocol for a hybrid type 1 randomized effectiveness-implementation trial using data science and economic incentive strategies to strengthen the continuity of care among people living with HIV in Tanzania. Trials. 2024 Feb 10;25(1):114. doi: 10.1186/s13063-024-07960-x. PMID 38336793
- [Derived] Kadota JL, Packel LJ, Mlowe M, Ulenga N, Mwenda N, Njau PF, Dow WH, Wang J, Sabasaba A, McCoy SI. Rudi Kundini, Pamoja Kundini (RKPK): study protocol for a hybrid type 1 randomized effectiveness-implementation trial using data science and economic incentive strategies to strengthen the continuity of care among people living with HIV in Tanzania. Res Sq [Preprint]. 2023 Dec 20:rs.3.rs-3315136. doi: 10.21203/rs.3.rs-3315136/v1. PMID 38196655